CLINICAL TRIAL: NCT04791566
Title: The Effects of Preoperative High-dose Dexamethasone on Inflammatory Response and Recovery After Emergency Laparotomy, a Randomized, Double-blind, Placebo-controlled Clinical Trial - AHA STEROID TRIAL
Brief Title: Preoperative High-dose Dexamethasone and Emergency Laparotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mirjana Cihoric (Other)
Responsible Party: Sponsor-Investigator, Mirjana Cihoric, MD, Research fellow, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-20038432
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Intestinal Obstruction and Ileus; Perforated Viscus; Sepsis; Pathophysiology; Inflammatory Response
MeSH Terms: conditions — Intestinal Obstruction; Ileus; Sepsis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intestinal obstruction, Dexamethasone 1 mg/kg (Active Comparator): Dexamethasone 1 mg/kg administered preoperatively as an i.v. infusion over 10-15 minutes
  Interventions: Drug: Dexamethasone 1 mg/kg
- Intestinal obstruction, PLACEBO (Placebo Comparator): Physiologic saline, administered preoperatively as an i.v. infusion over 10-15 minutes
  Interventions: Drug: Physiologic saline
- Perforated viscus, Dexamethasone 1 mg/kg (Active Comparator): Dexamethasone 1 mg/kg administered preoperatively as an i.v. infusion over 10-15 minutes
  Interventions: Drug: Dexamethasone 1 mg/kg
- Perforated viscus, PLACEBO (Placebo Comparator): Physiologic saline, administered preoperatively as an i.v. infusion over 10-15 minutes
  Interventions: Drug: Physiologic saline

INTERVENTIONS:
Drug: Dexamethasone 1 mg/kg — Dexamethasone 1 mg/kg administered as a single preoperative i.v. infusion over 10-15 min prior to general anaesthesia
  Other Names: Dexa-ratiopharm
  Arms: Intestinal obstruction, Dexamethasone 1 mg/kg; Perforated viscus, Dexamethasone 1 mg/kg
Drug: Physiologic saline — 100 mL Physiologic saline administered as a single preoperative i.v., infusion over 10-15 min prior to general anaesthesia
  Arms: Intestinal obstruction, PLACEBO; Perforated viscus, PLACEBO

SUMMARY:
The aim of this trial is to evaluate the effect of high-dose glucocorticoid on inflammatory response and recovery after emergency laparotomy in participants with intestinal obstruction and perforated viscus.

Primary outcome is the reduction of C-reactive protein on postoperative day 1. Secondary outcomes are organ specific complications in the post anaesthesia phase, endothel and inflammatory markers, fluid status, preload dependency, pain, lung function, nausea and mobilization during the first 5 days after surgery, .

The investigators hypothesize, that a preoperative single high dose of glucocorticoid reduces systemic inflammatory response after emergency laparotomy.

DETAILED DESCRIPTION:
Surgical trauma and accompanying inflammation results in increased capillary permeability leading to tissue edema. Since the vascular endothelium contributes to homeostasis, endothelial damage may increase the risk of cardiovascular and hemodynamic complications.

Pre-operative high-dose glucocorticoids provide reduction in the inflammatory response after surgery, effective pain relief in several major surgical procedures, as well as reducing fatigue, impairing endothelial dysfunction, potentially amend fluid extravasation, edema and dyscoagulation and vasodilation.

However, glucocorticoids have not been assessed in patients with peritonitis or intestinal obstruction, specifically, the impact on pain, fluid dynamics, respiratory as well as endothelial function and mobilization in both obstruction and perforation.

In this study, patients will be randomized to either high dose dexamethason (1 mg /kg) or placebo (0,9% NaCl), administered as a single dose preoperatively. The investigatoris hypothesize that a preoperative single high dose of glucocorticoid reduces systemic inflammatory response after emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years or over) undergoing emergency laparotomy (laparotomy or laparoscopy) for following abdominal pathology:

   1. Primary perforated viscus (perforated ulcer, small intestine or colon)
   2. Primary intestinal obstruction ( small intestine or colon)
2. Provided verbal and written informed consent
3. Must speak and understand the Danish language

Exclusion Criteria:

1. Appendectomies, cholecystectomies, negative diagnostic laparoscopies/laparotomies, herniotomies without bowel resections, sub-acute internal hernias after gastric bypass surgery, sub-acute surgery for inflammatory bowel diseases.
2. Emergency re-operations after elective surgery owing to paralytic/obstructive ileus, perforated viscus, anastomotic leakage
3. Reoperation owing to fascial separation with no other abdominal pathology identified and sub-acute colorectal cancer-surgery will be excluded from the cohort. Sub-acute surgery is defined as surgery planned within 48 hours.
4. Intestinal Ischemia
5. intraabdominal bleeding
6. Traumas, gynecological, urogenital and other vascular pathology, pregnant participants.
7. Dementia and/or cognitive dysfunction (diagnosed).
8. Participants not oriented in time, place and person
9. Insuline treatment for diabetes mellitus type I and II
10. Current treatment with systemic glucocorticoids or immune suppressive treatment ( apart from inhalation steroids)
11. Allergies to trial medicine

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
plasma C-reactive protein | 24* hours (*+/- 6 hours) after surgery.

SECONDARY OUTCOMES:
changes in plasma C-reactive protein | Preoperatively, 6 hours postoperatively, as well as postoperative day 3 and 5

OTHER OUTCOMES:
changes in postoperative inflammatory responses (IL-6, TNF alfa) | Preoperatively, 6 hours postoperatively, as well as postoperative day 1,3 and 5
Change in plasma Syndecain-1sE-Selectin (CD62E) | Preoperatively, 6 hours postoperatively, as well as postoperative day 1,3 and 5
Change in plasma soluble thrombomodulin (sTM)(CD141) | Preoperatively, 6 hours postoperatively, as well as postoperative day 1,3 and 5
Change in plasma sE-Selectin (CD62E) | Preoperatively, 6 hours postoperatively, as well as postoperative day 1,3 and 5
Change in vascular endothelial growth factor (VEGF) | Preoperatively, 6 hours postoperatively, as well as postoperative day 1,3 and 5
  0 to 1 point: Not high risk; 2 to 3 points: High risk
quick Sequential Organ Failure Assessment score, qSOFA | Assessed once preoperatively and 4 times daily during the first 5 postoperative days
Preload dependency via stroke volume(SV) guided resuscitation | Preoperatively, 6 hours postoperatively, as well as postoperative day 1,3 and 5
Fluid distribution, full body water via bioelectrical impedance vector analysis | Preoperatively, 6 hours postoperatively, as well as postoperative day 1,3 and 5
Peak flow measurements | Once a day on postoperative day 1,3 and 5
Postoperative need for antiemetic and analgesic beyond standard course | Once a day during the the first 5 postoperative days
Mobilization, The Cumulated Ambulation Score (CAS) | Once a day on postoperative day 1,3 and 5
  The CAS describes the patient's independence with regard to three activities (getting in and out of bed, sit-to-stand-to-sit from a chair, and walking). Each activity is assessed on a three-point ordinal scale from 0-2 (0 = Not able to, despite human assistance and verbal cueing, 1 = Able to, with human assistance and/or verbal cueing from one or more persons, 2 = Able to safely, without human assistance or verbal cueing, use of a walking aid allowed) resulting in a total daily CAS score ranging from zero to six
Postoperative delirium via Confusion Assessment method scale | Once a day during the the first 5 postoperative days
  1.a: Acute onset
  1b: Fluctuating course, 2: inattention 3: disorganized thinking 4: altered level of conciosness At least one criterion must be met for a positive result
Postoperative resting pain measured according to Numeric Rating Scale (NRS) | 6 hours after surgery as well as once a day one postoperative day 1,3 and 5
  0-10 where 0 is no pain and 10 is the worst pain imaginable
Postoperative pain during mobilization, measured according to Numeric Rating Scale (NRS) | 6 hours after surgery as well as once one postoperative day 1,3 and 5
  0-10 where 0 is no pain and 10 is the worst pain imaginable
30-day postoperative mortality | 30 days
90-day postoperative mortality | 90 days
30-day postoperative complications | 30 days
Length of ICU stay | 30 days
Overall hospital stay | 30 days
Plasma NO-bioavailability (L-arginine, asymmetric dimethylarginine) | preoperatively, 6 hours after surgery as well as once one postoperative day 1,3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Bang Foss, Professor, Study Director — Dept. of Anaesthesiology and Intensive Care
Locations (1):
- Mirjana Cihoric, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cihoric M, Kehlet H, Lauritsen ML, Hojlund J, Kanstrup K, Karnsund S, Foss NB. Preoperative high dose of dexamethasone in emergency laparotomy: randomized clinical trial. Br J Surg. 2024 Jul 2;111(7):znae130. doi: 10.1093/bjs/znae130. PMID 39028763